CLINICAL TRIAL: NCT06991595
Title: Fertility Limiting Diseases of Pelvic Organs and Their Influence on Receptivity of Endometrial Cavity: Prospective Clinical Trial (REAdME)
Brief Title: Fertility Limiting Diseases of Pelvic Organs and Their Influence on Receptivity of Endometrial Cavity: Prospective Clinical Trial
Acronym: REAdME
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: NU 23-06-00327
Record Dates: First submitted 2023-12-03; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Adenomyosis; Fibroid Uterus; Endometriosis
Keywords: adenomyosis; cytoreductive resection; myomectomy; endometriosis; endometrial receptivity
MeSH Terms: conditions — Adenomyosis; Leiomyoma; Endometriosis | interventions — Uterine Myomectomy; Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- adenomyosis: This project is divided into two parts - laboratory and clinical. This study utilizes a prospective, controlled, non-randomized design. In this study 5 main groups of infertile patients will be studied:women with severe adenomyosis (AD), uterine fibroids (UF), deep infiltrating endometriosis (DE),minimal or mild endometriosis (ETRS) and controls with only male factor of infertility and no signs ofpreviously mentioned diseases (CTRL). The patients will be recruited, and samples collected during the first 3 years of the project.
  Interventions: Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis; Procedure: hysteroscopy
- uterine fibroid: This project is divided into two parts - laboratory and clinical. This study utilizes a prospective, controlled, non-randomized design. In this study 5 main groups of infertile patients will be studied:women with severe adenomyosis (AD), uterine fibroids (UF), deep infiltrating endometriosis (DE),minimal or mild endometriosis (ETRS) and controls with only male factor of infertility and no signs ofpreviously mentioned diseases (CTRL). The patients will be recruited, and samples collected during the first 3 years of the project.
  Interventions: Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis; Procedure: hysteroscopy
- deep infiltrating endometriosis: This project is divided into two parts - laboratory and clinical. This study utilizes a prospective, controlled, non-randomized design. In this study 5 main groups of infertile patients will be studied:women with severe adenomyosis (AD), uterine fibroids (UF), deep infiltrating endometriosis (DE),minimal or mild endometriosis (ETRS) and controls with only male factor of infertility and no signs ofpreviously mentioned diseases (CTRL). The patients will be recruited, and samples collected during the first 3 years of the project.
  Interventions: Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis; Procedure: hysteroscopy
- minimal or mild endometriosis: This project is divided into two parts - laboratory and clinical. This study utilizes a prospective, controlled, non-randomized design. In this study 5 main groups of infertile patients will be studied:women with severe adenomyosis (AD), uterine fibroids (UF), deep infiltrating endometriosis (DE),minimal or mild endometriosis (ETRS) and controls with only male factor of infertility and no signs ofpreviously mentioned diseases (CTRL). The patients will be recruited, and samples collected during the first 3 years of the project.
  Interventions: Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis; Procedure: hysteroscopy
- controls: This project is divided into two parts - laboratory and clinical. This study utilizes a prospective, controlled, non-randomized design. In this study 5 main groups of infertile patients will be studied:women with severe adenomyosis (AD), uterine fibroids (UF), deep infiltrating endometriosis (DE),minimal or mild endometriosis (ETRS) and controls with only male factor of infertility and no signs ofpreviously mentioned diseases (CTRL). The patients will be recruited, and samples collected during the first 3 years of the project.
  Interventions: Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis; Procedure: hysteroscopy

INTERVENTIONS:
Procedure: cytoreductive resection of adenomyosis, myomectomy, resection of endometriosis — All women chosen for the study will be divided into the groups (AD, UF, DE, ETRS, CTRL) based on the inclusion/exclusion criteria (Table 2).A meticulous concern will be dedicated to patients´ education on advantages and disadvantages (including the eventual risks) of surgical and conservative management of AD and UF. These patients will be allocated into surgical or conservative arm of the study based on their inclinations: either to fertility saving surgical procedure (FSS) with subsequent IVF, or directly to IVF. This phenomenon of the importance of patients´ preferences in controversial clinical situations is the usual part of the management of infertile patients with AD or UF.
Procedure: hysteroscopy — Sampling of endometrium (Hysteroscopy) The samples will be collected using hysteroscopy, scheduled into the secretory phase of endometrial cycle. During hysteroscopy, the uterine cavity will be observed and described in the surgical protocol (capacity, symmetry, presence of intrauterine pathologies, internal ostia of the tubes). The 3.2 mm wide hysteroscope will be used. Its usage usually does not require any anaesthesia. The endometrium will be taken using biopsy forceps (7 French / 2.3 mm) and immediately frozen on dry ice and stored at -80 °C until processing. Two pieces of endometrium per patient will be collected - one for isolation of RNA and bulk RNA-Seq and/or RT-qPCR and the second one for isolation of nuclei and snRNA-Seq or validation using snRT-qPCR. If some unexpected findings would be observed during hysteroscopy (especially some interfering with fertility), they would be hysteroscopically removed and endometrial sampling postponed.

SUMMARY:
In this project, we will characterize the effects of fertility limiting diseases of pelvic organs on the receptivity of the endometrium. The primary aim of the project is the characterization of endometrium in patients with infertility suffering from AD, UF and DE, and compare it with infertile patients with minimal or mild endometriosis but no AD or UF (ETRS group), and with healthy women with only male factor of infertility (CTRL group, controls). The proper infertility treatment of patients with AD,UF and endometriosis is controversial and lacking clear evidence based algorithms. Despite their topical character, especially AD and DE (and UFs as well if present as multiple lesions) can be classified as systemic diseases in relation to women´s fertility. The presumed impact of these pathologies to endometrial receptivity (no matter they do not occur in the uterine cavity itself) can beseen as a fascinating hypothesis. Eradication of these diseases could have a potential to increase the prognosis of these women fundamentally.

DETAILED DESCRIPTION:
The project will be studied in two parts - laboratory and clinical. In the laboratory part, the parameters of endometrial receptivity will be specified in women with UF, AD, DE, minimal and mild endometriosis and in healthy controls. These parameters will be also compared in surgically treated patients before and after the procedures. This data will also be compared with patients from both control groups (ETRS, CTRL). First, we will perform bulk RNA Sequencing (RNA-Seq), to characterize the main differences in RNA expression of the endometrium between women with successful and unsuccessful conceptions. The candidate genes will be used for choosing the RTqPCR controlled set of samples for single-nucleus RNA-Seq (snRNA-Seq) profiling of the endometrial tissue. The results will be validated using RT-qPCR. In the clinical part, we will analyse the reproductive results of surgical and conservative management of infertility associated with AD and UF. Collectively, our data will provide information for the development of new diagnostic tools for better investigation and choice of treatment for patients with infertility. This project is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* agreement with participation in the study
* age between 18 - 45 years (at the start of patient´s participation in the study)women with at least 1 year infertility

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18-45 years
Study Population: * confirmed adenomyosis, score 3 or 4 [24]
  * planned conception using IVFwomen with at least 1 year infertility
  * confirmed uterine myoma/s with largest diameter from 25 to 55 mm and no interaction with uterine cavity (on US and hysteroscopy), i.e. types 3, 4, 5 or 6 [25]
  * presence of typical US features of leiomyomas [24]
  * planned conception using IVF women with typical symptoms of DE
  * confirmed DE (expert ultrasound and/or MRI) patients with confirmed endometriosis of stage I-II based on r-AFS [26]
  * planned conception patients without diseases mentioned above and with male factor of infertility
  * planned conception
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
loss of endometrial receptivity | 12 weeks
  frequency of patients with loss of receptivity

SECONDARY OUTCOMES:
pregnancy rate | 2 years
  the percentage of all attempts that leads to pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mara, Principal Investigator — General Hospital in Prague
Locations (1):
- General Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided